CLINICAL TRIAL: NCT07048015
Title: Effect of Hot Water Foot Bath on Daily Living Activities, Insomnia and Fatigue Levels in Frail Geriatric Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Munevver Kiyak, Nurse, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KGBSABGUYE
Record Dates: First submitted 2025-05-21; First posted 2025-07-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Frail Elderly
Keywords: frail elderly; foot bath; daily living activities; insomnia; fatigue; pain
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue; Pain

STUDY DESIGN:
Intervention Model Description: The first assessments (day 1) were made by the researcher using the Individual Identification Form, Katz Activities of Daily Living Scale, Insomnia Severity Index and Fatigue Severity Scale from patient files and face-to-face interviews with the patients. Foot bath was applied to the patients in the intervention group for 20 minutes once a day for 10 days. No intervention was made to the patients in the control group other than the medical treatment and care protocol. The second assessment was made on the 11th day by applying the , Katz Activities of Daily Living Scale, Insomnia Severity Index and Fatigue Severity Scale to the patients in the study and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foot bath (Experimental): Foot bath: The foot bath was applied to the patients in the intervention group once a day for 20 minutes for 10 days.
  Interventions: Other: Hot Water Foot Bath
- control group (No Intervention): No intervention was made to the patients in the control group other than the medical treatment and care protocol.

INTERVENTIONS:
Other: Hot Water Foot Bath — Hot Water Foot Bath:When the water temperature reached 40 ° C, the elderly person's feet were placed in the foot bath tub. The elderly person's feet were kept in the water for 20 minutes.
  Arms: Foot bath

SUMMARY:
Aim: A randomized controlled experimental study was conducted to determine the effect of hot water foot bath on daily living activities, sleep and fatigue levels in frail geriatric individuals.

Method: The study was conducted at Eskişehir Çifteler State Hospital internal medicine clinic between 15.10.2023 - 15.07.2024. 30 patients who met the sample selection criteria were randomized into two groups (study and control). Foot bath was applied to the study group every evening for 10 days. The study group was evaluated twice times on the 1st, 11th days, and the control group was evaluated twice on the 1st and 11th days in terms of frailty level, daily living activities, insomnia and fatigue severity.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and over
* At least literate
* Able to communicate
* With an Edmonton Frailty Scale score of 7 and above were included in the study.

Exclusion Criteria:

* Patients diagnosed with a disease that may affect their mental status, such as dementia
* Those who have used other treatment methods such as massage or cupping therapy in the last month
* Those whose systolic blood pressure is lower than 100 mmHg
* Those diagnosed with malignancy and acute inflammatory rheumatic disease
* Those who have undergone any surgical operation in at least 6 months
* Those who have an orthopedic implant (in the foot or leg area)
* Those who have paralysis and paralysis
* Those who have peripheral vascular disease
* Those who have ulcerative lesions in the legs
* Those who have a psychiatric disease diagnosis
* Those who are immobile
* Those who have fungal infections in their feet
* Those who are included in another study
* Those who have had a change in their treatment and nursing care process
* Those who have a diagnosis of neuropathy
* Patients who are allergic or sensitive to heat

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Effect of hot water foot bath on daily living activities, sleep and fatigue levels in frail geriatric individuals | from registration until the end of the 40th day
  Frail geriatric individuals were given hot water foot baths. The effects of this application on the individuals' daily living activities, sleep and fatigue levels were investigated. In the study, the individuals were administered the Edmoton Frailty Scale, the Katz Daily Living Activities Scale, the Insomnia Severity Index and the Fatigue Severity Scale via face-to-face interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malarvizhi, K. R. (2019). A study to assess the effectiveness of hot water foot bath therapy on quality of sleep among elderly staying in selected old age home at Villupuram District, Tamilnadu. International Journal of Health Sciences and Research, 4(4), 83-88.